CLINICAL TRIAL: NCT03330600
Title: Efficacy of Aquatic Physiotherapy in Stress Level and Muscle Tone of Children Between 3 and 24 Months With Microcephaly by Zika Virus Congenital Syndrome
Brief Title: Efficacy of Aquatic Physiotherapy in Children With Microcephaly by Zika Virus Congenital Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal de Pernambuco (Other)
Responsible Party: Principal Investigator, Milena Guimarães Monteiro, Principal investigator, Universidade Federal de Pernambuco
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: Projeto Milena LEPed
Record Dates: First submitted 2017-10-16; First posted 2017-11-06 (Actual); Last update posted 2019-05-07 (Actual); Status verified 2019-05

CONDITIONS: Zika Virus Infection; Microcephaly
MeSH Terms: conditions — Zika Virus Infection; Microcephaly | interventions — Hydrotherapy; Immersion

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- aquatic physicotherapy group (Experimental): For the experimental group, we will associate kinesiotherapy with immersion in water.
  Interventions: Behavioral: aquatic physicotherapy; Behavioral: immersion
- immersion group (Placebo Comparator): The control group will be submitted to immersion in the water, contained in flexion with the towel and maintaining the same care as the experimental one.
  Interventions: Behavioral: aquatic physicotherapy; Behavioral: immersion

INTERVENTIONS:
Behavioral: aquatic physicotherapy — Aquatic physiotherapy will be performed in a bathtub with water heated to a temperature around 37º C and environment with adequate temperature and luminosity. Kinesiotherapy will begin with smooth sliding movements in the aquatic environment, still in flexor restraint, allowing the child to adapt to the temperature of the new environment; joint mobilizations will be initiated on the shoulders and hips followed by stretching of the accessory muscles of the breath, spine erector, flexor and extensors of shoulder, elbow, hip, knee and ankle. The sessions will last 10 minutes and may be interrupted if the child shows signs of discomfort such as cyanosis, increased respiratory rate, bronchoaspiration or does not adapt to the environment, ie, remain crying for more than 5 minutes.
  Other Names: hydrotherapy
Behavioral: immersion — The immersion will be performed in a bathtub with water heated to a temperature around 37º C and environment with adequate temperature and luminosity. The therapy will begin with smooth sliding movements in the aquatic environment, still in flexor restraint, allowing the child to adapt to the temperature of the new environment. The sessions will last 10 minutes and may be interrupted if the child shows signs of discomfort such as cyanosis, increased respiratory rate, bronchoaspiration or does not adapt to the environment, ie, remain crying for more than 5 minutes.
  Other Names: hydrotherapy

SUMMARY:
Microcephaly associated with Congenital Syndrome of the Zika virus (SCVZ) was highlighted due to atypical structural and behavioral changes of the central nervous system. Such changes contribute to the appearance of functional impairments and difficulties of adaptation of the child to the necessary therapeutic follow-up. In this context, the search for adjuvant therapies that allow better management of these alterations has grown and, given its advantages, aquatic physiotherapy may be an auxiliary resource in the care of this population. The aquatic environment is capable of promoting a state of relaxation that, when associated with a kinesiotherapy protocol, is believed to have this potentiated effect. Thus, our objective will be to evaluate the efficacy of aquatic physiotherapy on the level of stress and muscle tone in children with microcephaly associated with SCVZ. A crossover, randomized, controlled and blind study will be carried out with children between 3 and 24 months of age, who will undergo two interventions: aquatic physiotherapy and water immersion. The evaluation of muscle tone will be performed through the Tardieu scale before and after the intervention; the physiological parameters (heart and respiratory rate, oxygen saturation and temperature) and the stress level will be evaluated before, immediately after and 30 minutes after the intervention. In addition, questionnaires will assess the child's behavioral state, level of irritation and sleep characteristics. For data normalization the Shapiro Wilk Test will be applied; the percentage values and relative frequency will be used for the descriptive analysis and for the numerical variables the values of mean and standard deviation or median and interquartile range. The paired T and ANOVA tests for repeated samples will be applied, which will analyze the intra-group time factor for the dependent variables of each individual. And for intergroup analysis, the variables may be submitted to the T-Test for independent or Mann-Whitney samples.

DETAILED DESCRIPTION:
A randomized, controlled, blind crossover study will be conducted at the Laboratory of Pediatric Studies (LEPED) located in the Physiotherapy Department of the Federal University of Pernambuco (UFPE), from January 2017 to November 2017. The study will be composed infants diagnosed with microcephaly associated with Zika virus Syndrome of the state of Pernambuco (PE), recruited for convenience of both sexes, aged 3 to 24 months of life.

Initially randomization of these children will be performed through randomization.com. and allocation in two groups (experimental and control) for the first session. After a period of one week (washout period), the groups are reversed so that everyone receives both interventions. Children in the experimental group will be submitted to a session of aquatic physiotherapy and the group control the immersion in water, described later. The study will be composed of two main researchers, the researcher 1 responsible for the intervention and the researcher 2 responsible for the evaluations, who will be blind to the intervention.

The collection of the clinical and sociodemographic data of the responsible person and the child will be done through the evaluation form developed for the research. Before the intervention, the child and the caregiver will be accommodated in a room with temperature, luminosity and controlled noises so that they can rest and thus minimize the effects of the route to the place of data collection. The evaluation begins with the assessment of muscle tone of the upper limbs and lower limbs, physiological parameters, postaral evaluation and application of questionnaires about maternal perception about the behavior of the and the level of stress. Immediately after the intervention will be reassessed muscle tone, physiological parameters and applied a questionnaire of maternal satisfaction about the therapy applied and perception of stress level.

ELIGIBILITY:
Inclusion Criteria:

* Infants aged 3 to 24 months, diagnosed with microcephaly according to the recommendations of the Surveillance Protocol and response to the occurrence of microcephaly and / or CNS disorders, which considers head circumference less than or equal to 31.5 cm for term boys and 31.9 cm for full term girls. In cases of prematurity, the perimeter will be considered less than 2 or more standard deviations according to the Intergrowth table for gestational age and sex. Mothers should report presence of skin rash or confirmation of Zika virus infection during pregnancy.
* Only children who are accompanied by a neurologist and assisted by physical therapy at least once a week will be included.

Exclusion Criteria:

* Children who are not taking anticonvulsant and / or antireflux medication when in the presence of seizures and gastroesophageal reflux, respectively;
* Infants who have less than 3 months of botulinum toxin application;
* Infants with osteomioarticular disorders, such as arthrogryposis, or other situations that impede the performance of evaluations and intervention;
* Children who are already active in the aquatic environment (hot tub or hydrotherapy).

Ages: 3 Months to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2018-02-18 (Actual); Study Completion 2018-10-30 (Actual)

PRIMARY OUTCOMES:
change in Modified Tardieu Scale | baseline and up 30 minutes
  assessment muscle tone at 5 degrees (0 = no resistance, 1 = slight resistance, no specific angle, 2 = moderate resistance with specific reaction angle, 3 = light clone, for less than 10 seconds, 4 = clusions for more than 10 seconds, 5 = immobile articulation). In addition to measuring the increase or decrease in the range of motion of each joint.

SECONDARY OUTCOMES:
change in heart rate | baseline and up 30 minutes
  rate of the heart's beat, recorded as the number of beats per minute.
change in respiratory frequency | baseline and up 30 minutes
  The number of breaths per minute.
change in oxygen saturation | baseline and up 30 minutes
  the fraction of the hemoglobin molecules in a blood sample that are saturated with oxygen at a given partial pressure of oxygen. Normal saturation is 95% to 100%.
change in body temperature | baseline and up 30 minutes
  the degree of sensible heat or cold, expressed in terms of Celsius

CONTACTS AND LOCATIONS:
Overall Officials: Karla Mônica Ferraz Lambertz, Study Chair — Universidade Federal de Pernambuco
Locations (1):
- Universidade Federal de Pernambuco, Recife, Pernambuco, Brazil

IPD SHARING:
Plan to Share IPD: No